CLINICAL TRIAL: NCT03907800
Title: Neoadjuvant Nab-paclitaxel in Triple-negative or HER2-positive Breast Cancer
Acronym: NeoPATH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Li Zhu, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1801
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Carboplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel + Carboplatin ± Herceptin (Experimental)
  Interventions: Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Herceptin

INTERVENTIONS:
Drug: Nab-paclitaxel — 125 mg/m² weekly, infusion, 3 weeks on 1 week off, applicated for four cycles.
Drug: Carboplatin — AUC 2, weekly, 3 weeks on 1 week off, applicated for 4 cycles
Drug: Herceptin — In case of HER2-positive, patients receive Herceptin weekly during all cycles.

SUMMARY:
To evaluate the efficacy and safety of nab-paclitaxel combined with carboplatin for Chinese patients with triple-negative and HER2-positive breast cancer in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study according to local regulatory requirements prior to beginning specific protocol procedures.
2. Age at diagnosis ≥ 18 years, female.
3. Histologically confirmed diagnosis of HER2-opsitive or triple-negative breast cancer. ER/PR-negativity is defined as ≤1% stained cells； HER2-positivity is defined as IHC 3+ or in-situ hybridisation (ISH) ratio >2.0.
4. cT2-4NanyM0 or cTanyN1-3M0
5. ECOG ≤ 1, LVEF ≥ 55%.
6. Laboratory requirements: for hematology, absolute neutrophil count (ANC) ≥ 1.5 × 109 / L and platelets ≥ 100 × 109 / L and hemoglobin ≥ 90 g/L; for hepatic function, total bilirubin ≤ 1.5 × UNL, AST and ALT ≤ 2.5 × UNL; for renal function, SCr ≤ 1.5 × UNL
7. Patients must be available and compliant for treatment and follow-up.

Exclusion Criteria:

1. Prior chemotherapy, endocrine therapy or radiation therapy for any malignancy.
2. Known or suspected congestive heart failure (> NYHA I)
3. Currently active infection or severe symptomatic visceral disease.
4. Definite contraindications for the use of corticosteroids or known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol
5. rior malignancy with a disease-free survival of < 5 years, except curatively treated basalioma of the skin, pTis of the cervix uteri.
6. Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
7. Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (ypT0/is ypN0) rate | 16 weeks (at the time of definitive surgery)
  Absence of invasive cancer in the breast and axillary nodes, irrespective of ductal carcinoma in situ.

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) | 5 years
  IDFS is defined as the time period between registration and first event (ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, second primary nonbreast invasive cancer)
Distant disease-free survival (DDFS) | 5 years
  DDFS is defined as the time period between registration and first event (distant recurrence, death attributable to any cause, second primary nonbreast invasive cancer)
Objective response rate (ORR) | 16 weeks (at the time of definitive surgery)
  ORR includes all patients whose cancer has a partial or complete response according to RECIST 1.1
Breast conservation rate | 16 weeks (at the time of definitive surgery)
  To determine the breast conservation rate after neoadjuvant treatment.
Tolerability and safety: number of patients whose treatment had to be reduced, delayed or permanently stopped | during treatment (16 weeks)
  Descriptive statistics will be given on the number of patients whose treatment had to be reduced, delayed or permanently stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhu, Prof., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD